# Correlation of Audiovisual Features With Clinical Variables and Neurocognitive Functions in Bipolar Disorder, Mania

01.08.2017

# **Statistical Analysis**

# **Speech and Video Analysis**

Classification Methods

Feature vectors extracted from audio and video are modelled using Partial Least Squares (PLS) regression and Extreme Learning Machines based classifiers (Kaya et al., 2015; 2017).

### **Neurocognitive Evaulation**

Statistical evaluation is done by using SPSS(Statistical Package for Social Sciences) for Windows 18.0 program. Categoric variables are compared with Chi-square test, qualitative variables are compared with dependent and independent sampling t-test and Mann- Whitney U test. Correlation analysis are done with Pearson and Spearman test. Statistical significance is \*=p<0.05, \*\*=p<0.01, all of tests are two-sided.

# Emotion predictions for Pearson correlation analysis and regression of YMRS drop

# Regression Model

YMRS score temporal change is calculated as, t1=0th day, t2=3rd day, t3=7th day, t4=14th day, t5= 28th day, t6=90th day and X1=t2/t1, X2=t3/t1, X3=t4/t1, X4=t5/t1 and X5=t6/t1. These proportions are regressed as stepwise linearly to valence, arousal and singular affect scores of first audio recording values.